CLINICAL TRIAL: NCT05007223
Title: Characterization and Analysis of the Skin Microbiome in Hailey-Hailey Disease
Brief Title: Skin Microbiome Profile in Hailey-Hailey Disease
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sang Eun Lee, Assistant professor, Gangnam Severance Hospital
Other Study IDs: 3-2020-0106
Record Dates: First submitted 2021-08-05; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Hailey-Hailey Disease
MeSH Terms: conditions — Pemphigus, Benign Familial | interventions — Doxycycline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Case (HHD) 1) Axillar active lesion 2) Axillar healed lesion 3) Inguinal active lesion 4) Inguinal healed lesion
  2. Control (NC) 1) Axillar area 2) Inguinal area
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1. Experimental: doxycycline: Given doxycycline and assessment of skin
  Interventions: Drug: Doxycycline
- 2. No Intervention: Healthy Controls: Control subjects to assess if there is baseline difference in the skin microbiome

INTERVENTIONS:
Drug: Doxycycline — 200mg/day for 28 days(Given doxycycline to patients with Hailey-Hailey disease)
  Groups: 1. Experimental: doxycycline

SUMMARY:
"Hailey-Hailey disease is an autosomal dominant disorder caused by a genetic defect in a calcium ATPase (ATP2C1) leading to a defect in keratinocyte adhesion. The characteristic of this disease is the involvement of intertriginous areas of the skin, which are the moist sites including the axillary vault and the inguinal crease. The composition of microbial communities is primarily dependent on the physiology of the skin site and the moist sites have distinct compositions of skin microorganisms. In addition, treatment with doxycycline is often helpful in the management of Hailey-Hailey disease. These findings suggest a role of the skin microbiome in the pathogenesis of Hailey-Hailey disease.

The purpose of this study is to characterize the skin microbiome in patients with Hailey-Hailey disease by the 16S method, to better understand the pathogenesis of the disease and to discover new therapeutic targets in the future.

DETAILED DESCRIPTION:
Investigators will look at patients with Hailey-Hailey disease, and healthy controls.

Investigators will look at skin microbiome (Bacterial diversity and the relative abundance of major bacterial taxa) Investigators will assess this in patients with Hailey-Hailey disease before and after doxycycline and compare them to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. Hailey-Hailey disease 1-1. Inclusion Criteria

1. Clinically diagnosed with Hailey-Hailey as confirmed by histopathology and/or genetic analysis.
2. >19 years old
3. Patients who currently have lesions on the axilla and groin
4. Patietns who signed the consent form and Informed Consent in Human Material Research

2. Normal control 2-1. Inclusion Criteria

1. >19 years old
2. Persions who signed the consent form and Informed Consent in Human Material Research

Exclusion Criteria:

1-2. Exclusion Criteria

1. Patients who have used systemic steroids or antibiotics within the last 1 month
2. Patients who have used local steroids or antibiotics within the last 2 weeks
3. Patients who have been diagnosed with skin diseases(such as atopic dermatitis) other than Hailey-Hailey disease
4. Patients who are unable to swab or who may have affect a medical condition
5. Patients who have difficulty making clear decisions due to lack of decision-making ability
6. In addition to the above, a person who is considered inappropriate to participate in this study, such as collecting test information, based on the medical judgment of the Principal investigator or Subinvestigator.

2-2. Exclusion Criteria

1. Persions who have skin diseases(such as atopic dermatitis) or diseases affecting the skin microbes
2. Persions who have used systemic steroids or antibiotics within the last 1 month
3. Patients who have used local steroids or antibiotics within the last 2 weeks
4. In addition to the above, a person who is considered inappropriate to participate in this study, such as collecting test information, based on the medical judgment of the Principal investigator or Subinvestigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Hailey Hailey, diagnosis confirmed by histopathology or genetics at Gangnam Severance Hospital, Dermatology Department
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Shannon diversity index | 1 year
  1. Change in the bacterial diversity index of the skin microbiome in those with and without Hailey-Hailey disease.
  2. Change in the bacterial diversity index of the skin microbiome before and after the treatment of doxycycline in those with Hailey-Hailey disease
  The diversity will be evaluated by assessing the Shannon diversity of the bacterial DNA in the skin microbiome

SECONDARY OUTCOMES:
OTU(Operational Taxonomic Unit) | 1 year
  1. Change in the relative abundance of major bacterial taxa of skin microbiome in those with and without Hailey-Hailey disease
  2. Change in the relative abundance of major bacterial taxa of skin microbiome before and after the treatment of doxycycline in those with Hailey-Hailey disease
  The representative Operational Taxonomic Unit (OTU) sequences were assigned to a taxonomy at a confidence threshold of 50% using remote desktop protocol classifier with reference to the Greengenes database. Relative abundance of OTUs based on all unique sequences was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Eun Lee, Principal Investigator — Department of Dermatology, Gangnam Severance Hospital, Yonsei University College of Medicine,
Locations (1):
- GangnamSeveracne Hospital, Seoul, South Korea